CLINICAL TRIAL: NCT00360685
Title: Safety of Tacrolimus And Methotrexate (MTX) Versus Tacrolimus And Mycophenolate Mofetil (MMF) As Graft Versus Host Disease Prophylaxis In Allogeneic Hematopoietic Cell Transplants (HCT)
Brief Title: Tacrolimus and Mycophenolate Mofetil (MMF) in GVHD Prophylactic Regimen Compared to Tacrolimus and Methotrexate (MTX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-14418
Record Dates: First submitted 2006-08-03; First posted 2006-08-07 (Estimated); Results first posted 2013-05-03 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-03

CONDITIONS: Mucositis; Graft-versus-host Disease
Keywords: Tacrolimus; Methotrexate; Mycophenolate mofetil; Mucositis; Acute graft-versus-host disease (aGVHD); Engraftment; hemolytic/uremic syndrome (HUS); Thrombotic thrombocytopenic purpura (TTP)
MeSH Terms: conditions — Mucositis; Graft vs Host Disease; Hemolytic-Uremic Syndrome; Purpura, Thrombotic Thrombocytopenic | interventions — Tacrolimus; Methotrexate; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAC + MMF (Other): Tacrolimus and Mycophenolate
  Interventions: Drug: TAC + MMF
- TAC+MTX (Other): Tacrolimus and Methotrexate
  Interventions: Drug: Tac+MTX

INTERVENTIONS:
Drug: Tac+MTX — Tacrolimus- 0.03mg/kg/24h IV beginning day-3 Methotrexate- 15mg/m2 IV day +1 then 10mg/m2 IV on days 3, 6, 11 post transplant.
  Other Names: Tacrolimus, Prograf(R); Methotrexate,
  Arms: TAC+MTX
Drug: TAC + MMF — Tacrolimus- 0.03 mg/kg/24h as a continuous IV infusion, beginning day -3. Mycophenolate Mofetil- 30 mg/kg/day IV in 2 divided doses (q12 hours) beginning day 0 at least 2 hours after the end of the hematopoietic stem cell transplant
  Other Names: Tacrolimus, Prograf(R); Mycophenolate mofetil, CellCept(R)
  Arms: TAC + MMF

SUMMARY:
A comparative trial where all patients will receive daily doses of tacrolimus (TAC) until day +60 when tapering will begin, in the absence of graft-versus-host disease (GVHD), and discontinued by day +180. In addition patients will be randomized to methotrexate (MTX) or mycophenolate mofetil (MMF) and again, in the absence of GVHD, a tapering schedule will begin on day +240 and be completed on day +360. Doses will be adjusted to maintain blood levels.

DETAILED DESCRIPTION:
The randomization for this comparative trial will be stratified by conditioning regimen and, for those patients enrolled on MCC-14178, by busulfan AUC level.

All patients will receive daily doses of TAC beginning day -3 (day 0 being the day of hematopoietic stem cell transplant (HCT)) and will be given until day +60 when tapering will begin in the absence of GVHD. Provided no GVHD develops, TAC should be discontinued by day +180. Doses will be adjusted to maintain blood levels.

In addition to TAC, patients will be randomized to one of the following additional anti-GVHD medications: MTX or MMF beginning day 0 at least 2 hours after the end of the HCT. In the absence of GVHD a tapering schedule will begin on day +240 and be completed on day +360.

Study participants will be extensively monitored as inpatients and then weekly as outpatients. Some tests will be conducted at least twice weekly (blood tests, toxicity data, GVHD and physical exams) one-month post-transplant and during the tapering off periods for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

- Patient must be going through a T cell-replete allogeneic transplant

Exclusion Criteria:

- A contraindication to the use of tacrolimus, mycophenolate, or methotrexate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2005-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janelle Perkins, PharmD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute; Teresa Field, PhD, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States

REFERENCES:
- [Background] Perkins J, Field T, Kim J, Kharfan-Dabaja MA, Fernandez H, Ayala E, Perez L, Xu M, Alsina M, Ochoa L, Sullivan D, Janssen W, Anasetti C. A randomized phase II trial comparing tacrolimus and mycophenolate mofetil to tacrolimus and methotrexate for acute graft-versus-host disease prophylaxis. Biol Blood Marrow Transplant. 2010 Jul;16(7):937-47. doi: 10.1016/j.bbmt.2010.01.010. Epub 2010 Jan 25. PMID 20102746
- See also: Moffiitt Cancer Center Clinical Trials Website — http://www.moffitt.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Tacrolimus And Methotrexate: All patients will receive TAC 0.03 mg/kg/24h as a continuous IV infusion beginning day -3 (day 0 being the anticipated day of hematopoietic stem cell infusion). Tacrolimus dosing should be based on ideal body weight. TAC levels should be measured on day 0 then at least twice weekly for the first month and the dose will be adjusted to maintain whole blood levels of 5-15ng/mL. When the patient is able to tolerate oral medications, the total daily dose of IV TAC will be converted to oral dosing at a 1:3 (IV:PO) ratio. The daily oral dose will be divided into twice daily dosing. Full dose TAC will be given until day +60 (+7) when tapering will begin in the absence of GVHD. Provided no GVHD develops, TAC should be discontinued by day +180 (+14).
  MTX 15 mg/m2 IV day +1 then 10 mg/m2 IV on days +3, +6, and +11.
- Tacrolimus And Mycophenolate Mofetil: All patients will receive TAC 0.03 mg/kg/24h as a continuous IV infusion beginning day -3. TAC levels should be measured on day 0 then at least twice weekly for the first month and the dose will be adjusted to maintain whole blood levels of 5-15ng/mL. When the patient is able to tolerate oral medications, the total daily dose of IV TAC will be converted to oral dosing. Full dose TAC will be given until day +60 (+7) when tapering will begin in the absence of GVHD. Provided no GVHD develops, TAC should be discontinued by day +180 (+14).
  MMF 30 mg/kg/day IV in 2 divided doses beginning day 0. Dosing should be based on the lesser of adjusted ideal body weight or actual body weight. The IV dose will be converted to the oral formulation when spatient is able to tolerate oral medications. Oral dosing may be capped at 1 gram twice daily. In the absence of GVHD a tapering schedule will begin on day +240 (+14) and be completed on day +360 (+14).
Period: Overall Study
Arm/Group | Tacrolimus And Methotrexate | Tacrolimus And Mycophenolate Mofetil
Started | 47 | 42
Completed | 47 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Tacrolimus And Methotrexate: Tacrolimus (TAC) And Methotrexate (MTX)
- Tacrolimus And Mycophenolate Mofetil: Tacrolimus (TAC) And Mycophenolate Mofetil (MMF)
- Total: Total of all reporting groups
Arm/Group | Tacrolimus And Methotrexate | Tacrolimus And Mycophenolate Mofetil | Total
Number analyzed (Participants) | 47 | 42 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 39 | 84
  >=65 years | 2 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 21 | 39
  Male | 29 | 21 | 50
Region of Enrollment [Number; unit: participants]
  United States | 47 | 42 | 89

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Severe Mucositis
Description: Mucositis was assessed prospectively daily while the patient was hospitalized and graded retrospectively based on nurse and clinician assessments according to the clinical criteria set forth in the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE; version 3.0). Severe mucositis as defined as grade 3 or grade 4.
Time Frame: 2 year
Population: Intent to treat
Measure: Number; unit: participants
Groups:
- Tacrolimus And Methotrexate: Tacrolimus And Methotrexate
Arm/Group | Tacrolimus And Methotrexate | Tacrolimus And Mycophenolate Mofetil
Number analyzed (Participants) | 47 | 42
participants | 25 | 14
Statistical Analysis 1: Comparison: Tacrolimus And Methotrexate vs Tacrolimus And Mycophenolate Mofetil; Sample size was based on the difference in the proportion of patients in each arm who were predicted to develop severe mucositis defined as clinical grade 3 or 4 per the CTCAE. A sample-size of 42 evaluable subjects per study-arm allowed detection of an absolute difference of 30%, which corresponds to a reduction in the incidence of severe mucositis from 60% in the methotrexate arm to 30% in the MMF arm (alpha=0.05, power=0.80); Test type: Superiority or Other; p = 0.06, Fisher Exact

2. Secondary Outcome: Incidence of Acute Graft-vs-host Disease (aGVHD)
Description: incidence of aGVHD (grades 2 - 4) 100 days post allogeneic hematopoietic cell transplantation
Time Frame: 100 days post transplant
Population: intent to treat
Measure: Number; unit: participants
Arm/Group | Tacrolimus And Methotrexate | Tacrolimus And Mycophenolate Mofetil
Number analyzed (Participants) | 47 | 42
participants | 45 | 33
Statistical Analysis 1: Comparison: Tacrolimus And Methotrexate vs Tacrolimus And Mycophenolate Mofetil; Test type: Superiority or Other; p = 0.8, K-sample tests for comparing the cumulat

3. Secondary Outcome: Overall Survival
Description: number of participants alive at one year
Time Frame: 1 year
Population: intent to treat
Measure: Number; unit: participants
Arm/Group | Tacrolimus And Methotrexate | Tacrolimus And Mycophenolate Mofetil
Number analyzed (Participants) | 47 | 42
participants | 28 | 27
Statistical Analysis 1: Comparison: Tacrolimus And Methotrexate vs Tacrolimus And Mycophenolate Mofetil; Test type: Superiority or Other; p = 0.58, Log Rank

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Tacrolimus And Methotrexate | Tacrolimus And Mycophenolate Mofetil
Serious Adverse Events (participants affected / at risk) | 25/47 | 19/42
Other Adverse Events (participants affected / at risk) | 0/47 | 0/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tacrolimus And Methotrexate (N=47) | Tacrolimus And Mycophenolate Mofetil (N=42)
Death (General disorders) | 25 (25) | 19 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes